CLINICAL TRIAL: NCT05769348
Title: Investigation and Modulation of the Central Mu-Opioid Mechanism in Migraine (in Vivo)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Alexandre DaSilva, DDS, DMedSc, Director of the Headache and Orafacial Pain Effort Lab, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00213295; R01NS094413 (NIH)
Record Dates: First submitted 2023-02-13; First posted 2023-03-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will not know if they are receiving active or sham treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Active Unilateral Treatment (Active Comparator): Chronic migraine patients will be randomized (Taves method) to receive UNILATERAL high-definition transcranial direct current stimulation (HD-tDCS*) as 20 minute sessions, once daily for 20 days (M-F for 4 weeks).
  Interventions: Device: HD-tDCS Active Protocol
- Active Bilateral Treatment (Active Comparator): Chronic migraine patients will be randomized (Taves method) to receive BILATERAL high-definition transcranial direct current stimulation (HD-tDCS*) as 20 minute sessions, once daily for 20 days (M-F for 4 weeks).
  Interventions: Device: HD-tDCS Active Protocol
- Sham Treatment (Sham Comparator): Chronic migraine patients will be randomized (Taves method) to receive SHAM high-definition transcranial direct current stimulation (HD-tDCS*) as 30-second administrations at the beginning and end of each 20 minute session, once daily for 20 days (M-F for 4 weeks).
  Interventions: Device: HD-tDCS Sham Protocol
- No Treatment (No Intervention): Episodic Migraine Patients will not receive study treatment. These patients will complete observational study components (Screening visit, baseline visit, MRI and PET scan only).

INTERVENTIONS:
Device: HD-tDCS Active Protocol — non-invasive brain stimulation (active protocol)
  Arms: Active Bilateral Treatment; Active Unilateral Treatment
Device: HD-tDCS Sham Protocol — non-invasive brain stimulation (sham protocol)
  Arms: Sham Treatment

SUMMARY:
This study investigates whether unilateral and bilateral non-invasive brain stimulation, given for 20 minutes/once per day for twenty days (M-F) can reduce migraine pain. Fourty patients will receive treatment (20 unilateral treatment, and 20 bilateral treatment), while twenty will receive a "sham" procedure. Another 20 Episodic Migraine patients will be recruited for the observational aim of the study which does not include brain stimulation.

DETAILED DESCRIPTION:
Clinical Trial:

This is a phase 2, single center, three-arm, double-masked, randomized investigation and modulation of the µ-opioid and D2/D3 mechanisms in chronic migraine (in vivo). We will enroll 60 patients with Chronic Migraine divided into 3 Lab/Home-Based groups: 20 for the active unilateral M11-2 HD-tDCS group, 20 for the active bilateral M11-2 HD-tDCS group, and 20 for the sham M11-2 HD-tDCS group. Patients will complete a screening visit, baseline visit with MRI and PET session, 20 days of HD-tDCS brain stimulation treatments, as well as follow-up visits with an MRI and PET session.

Observational Study Arm:

20 additional patients with low frequency EM (<8 attacks/month) patients (that did not undergo neuromodulation) will be recruited for the study. Historical data may be used in place of recruiting new participants. Data from these 20 EM volunteers will be compared to that of CM patients at baseline; however, they will not be part of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 (inclusive)
* Patients must have Episodic migraines that started before the age of 50, and currently experience:

  * Chronic migraine (ICHD-3-beta), headache occurring on 15 days/month for more than six months, which, on at least eight days/month, has the features of a migraine headache.
  * Episodic migraine (low frequency), specifically those with headache occurring less than 8 days/month.
* Willing to limit the introduction of new treatments and medications during the study period.

Exclusion Criteria:

* Significantly greater pain in body sites other than the head
* Active, untreated major concurrent systemic illness other than migraine

  * Medical conditions that can impair health status independent of migraine (including cardiopulmonary disorders, malignancy, uncontrolled endocrine or allergies)
  * Systemic rheumatic disorders (i.e., rheumatoid arthritis, systemic lupus erythematosus, gout, and fibromyalgia);
* History or current evidence of a psychotic disorder (e.g., bipolar disorder, schizophrenia) or severe major depression, as evidenced by Beck Depression score of >30*
* History of neurological disorder (e.g., epilepsy, stroke, neuropathy, neuropathic pain)
* Medication overuse headache (ICHD-3), regular intake for ≥10 days per month of ergotamine, triptans, combination analgesics, or any combination thereof OR ≥15 days per month of simple analgesics (acetaminophen, aspirin, NSAID), for more than 3 months
* Current use of opioid or dopaminergic drugs (or use within the last 3 months) or substance abuse (self-reported)
* Drug test positive for opioid or recreational drug (e.g., cannabis) at the time of the PET scan visits
* Allergic response to study radiotracers or chemically related drugs
* Excluded by MRI Center or PET Center safety screening checklist (as administered by study staff)
* Pregnant or lactating (negative urine pregnancy test must be available before any PET procedures are initiated)
* Prior use of tDCS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in moderate to severe headache days over 1 month follow-up | baseline to 1 month follow-up
  Headache Day: day with a headache that causes moderate or severe pain (at its peak, defined as NRS ≥ 4) that lasts at least 4 hours, OR day with a headache that is treated by an acute headache medication.

SECONDARY OUTCOMES:
Change from baseline in headache days over 1-month follow-up | baseline to 1 month follow-up
  Day with a headache that lasts at least 2 hours, OR day with a headache that is treated by an acute headache medication.
Responder rate over 1-month follow-up | baseline to 1 month follow-up
  50% percent reduction (from baseline to post tDCS) in the number of moderate or severe headache days.
Changes from baseline in medication use days over 1-month follow-up | baseline to 1 month follow-up
  - Medication use is defined as a day when the patient reports intake of medication for the acute treatment of headache
Intensity of headache over 1-month follow-up | baseline to 1 month follow-up
  Each headache day is rated in terms of maximum intensity on a 0 to 10 NRS scale and averaged headache intensity will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre DaSilva, DDS, DMedSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No